CLINICAL TRIAL: NCT02818569
Title: Repurposing Dexmedetomidine as an Orally Administered Sleep Therapeutic
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Oluwaseun Johnson-Akeju, MD, MMSc, Assistant Professor in Anesthesia, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016P000269
Record Dates: First submitted 2016-06-13; First posted 2016-06-29 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Sleep; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will receive both the oral dexmedetomidine intervention and placebo comparator in a randomized order.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Dexmedetomidine, Then Placebo (Experimental): This arm will enroll healthy control subjects, who will have an acclimation night followed by a night's sleep with oral dexmedetomidine and then a night's sleep with a placebo comparator.
  Interventions: Drug: Dexmedetomidine; Other: Saline Placebo
- Placebo, Then Oral Dexmedetomidine (Experimental): This arm will enroll healthy control subjects, who will have an acclimation night followed by a night's sleep with a placebo comparator and then a night's sleep with oral dexmedetomidine .
  Interventions: Drug: Dexmedetomidine; Other: Saline Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Oral form
  Other Names: Precedex
Other: Saline Placebo — Saline Placebo
  Other Names: Saline

SUMMARY:
The broad objective of this investigation is to assess the safety and efficacy of oral therapy with dexmedetomidine for the induction and maintenance of restful sleep.

DETAILED DESCRIPTION:
Sleep is a basic human function that occupies approximately one-third of our lives. Much of what is known about the benefits of sleep in humans has been obtained from studies of patients with insomnia, the most common sleep disorder with a reported prevalence of 10 to 15%. Unfortunately, insomnia is an independent risk factor for acute myocardial infarction, coronary heart disease, heart failure, hypertension, diabetes, and death. More so, sleep disturbances lead to neurocognitive deficits such as delirium and psychosis. However, the principal medications (i.e. benzodiazepines, zolpidem) currently used to treat insomnia are associated with side effects such as daytime sedation, delirium, anterograde memory disturbance, and complex sleep-related behaviors. We recently found that a nighttime intravenous bolus administration of dexmedetomidine was associated with normal sleep architecture comprising of rapid eye movement (REM) and non-REM (N1, N2, N3) sleep, with improved next-day psychomotor vigilance performance compared to zolpidem. Presently, dexmedetomidine is only available in an intravenous formulation. The goal of this project is to develop dexmedetomidine, an alpha-2 receptor agonist, into an oral sleep therapeutic with a neurocognitive sparing profile.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-50
* Native English speaking
* ASA physical status classification P1 and P2 (stable chronic condition)
* Normal body habitus.

Exclusion Criteria:

* Abnormal sleep habits
* Sleeping less than 5 hours each night
* Going to sleep before 9:00 PM or after 2:00 AM on a regular basis
* Waking up before 5:00 AM or after 10:00 AM on a regular basis.
* Takes medication that alters sleep, cognitive function, or both. -Has a history of a known neurological or psychiatric problem.
* Younger than 18 or older than 50 years of age.
* Known or suspected sleep disorder(s).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are undecided.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 15 participants completed both arms (dexmedetomidine and placebo) for the study. After being randomized and completing the first arm, patients completed the alternative arm thereafter.
Groups:
- Placebo, Then Oral Dexmedetomidine: This arm will enroll healthy control subjects, who will have an acclimation night followed by a night's sleep with a placebo comparator and then a night's sleep with oral dexmedetomidine.
Period: Overall Study
Arm/Group | Oral Dexmedetomidine, Then Placebo | Placebo, Then Oral Dexmedetomidine
Started (All 15 patients were enrolled in both study arms, undergoing sleep with oral dex and a placebo.) | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All 15 Participants completed both arms of the study. After being randomized and completing a single arm, they proceeded to complete the second arm thereafter.
Groups:
- All Study Participants: All study participants who were either randomized to receive either Oral Dexmedetomidine or the placebo comparator initially.
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants] — Population: All 15 Participants completed both arms of the study. After being randomized and completing a single arm, they proceeded to complete the second arm thereafter.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 15
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All 15 Participants completed both arms of the study. After being randomized and completing a single arm, they proceeded to complete the second arm thereafter.
  Participants
    Female | 8
    Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All 15 Participants completed both arms of the study. After being randomized and completing a single arm, they proceeded to complete the second arm thereafter.
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 13
    Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All 15 Participants completed both arms of the study. After being randomized and completing a single arm, they proceeded to complete the second arm thereafter.
  Participants
    American Indian or Alaska Native | 0
    Asian | 6
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 8
    More than one race | 1
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Hemodynamic Stability (Phase I)
Description: Number of participants with (1) systolic blood pressure (SBP) < 60 mmHg, diastolic blood pressure (DBP) < 40 mmHg or decrease of SBP by ≥ 50 % from the baseline which is sustained over two consecutive minutes, (2) hypertension: SBP > 180 mmHg, DBP > 100 mmHg, or increase of SBP by ≥ 50 % from the baseline which is sustained over two minutes and, (3) bradycardia: heart rate (HR) < 40 bpm or decrease by ≥ 50 % from the baseline sustained over two consecutive minutes.
Time Frame: Active study night, visit 3 or 4
Measure: Count of Participants; unit: Participants
Groups:
- Oral Dexmedetomidine: Dexmedetomidine
  Type: Oral
- Placebo Comparator: Placebo Comparator
  Type: Saline
Arm/Group | Oral Dexmedetomidine | Placebo Comparator
Number analyzed (Participants) | 15 | 15
Participants
  SBP < 60 mmHG | 0 | 0
  Hypertension | 0 | 0
  Bradycardia | 0 | 0

2. Primary Outcome: Polysomnography Sleep Quality (Phase II).
Description: Number of participants who had EEG features of natural sleep. Relative quantities of spindles and k-complexes were used to assess approximation to natural sleep.
Time Frame: Active study night, visit 3 or 4
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- Oral Dexmedetomidine: Oral Dexmedetomidine
- Placebo Comparator: Saline
  Saline Placebo: Saline Placebo
Arm/Group | Oral Dexmedetomidine | Placebo Comparator
Number analyzed (Participants) | 15 | 15
participants | 15 | 15

3. Secondary Outcome: Performance on the Psychomotor Vigilance Task (Phase II)
Description: The number of responses that were longer than 400 milliseconds (lapse 400).
Time Frame: Active study night, visit 3 or 4
Measure: Mean (Standard Deviation); unit: lapses
Groups:
- Experimental: Oral Dexmedetomidine
  Dexmedetomidine: Oral form
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 15 | 15
lapses
  Training (Before Sleep) | 5.8 (5) | 6.5 (7)
  Testing (After Sleep) | 14.5 (15.5) | 12.3 (13.2)

4. Secondary Outcome: Performance on the Motor Sequence Task (Phase II)
Description: Number of participants with improved MST score after sleeping.
Time Frame: Active study night, visit 3 or 4
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 15 | 15
Participants | 12 | 13

5. Secondary Outcome: Subjective Sleep Quality (Phase II)
Description: Self-reported sleep latency.
Time Frame: Active study night, visit 3 or 4
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 15 | 15
minutes | 33 (24.4) | 36.3 (27.3)

ADVERSE EVENTS:
Time Frame: Length of study conduction through visits 1-4
Arm/Group | Experimental | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT02818569/Prot_SAP_000.pdf